CLINICAL TRIAL: NCT02079831
Title: Effects of Varied Macronutrient Composition on Weight Loss in Obese Adolescents
Brief Title: PrOtein and WEight Loss in teenageRs
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 2014-014
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Pediatric Obesity
Keywords: Adolescent obesity; childhood obesity; anthropometry; body weights and measures
MeSH Terms: conditions — Pediatric Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher protein and energy restriction (Experimental): Participants in this arm will consume 30% of energy as protein with 25% energy restriction.
  Interventions: Behavioral: Energy Restriction; Behavioral: Higher protein
- Lower protein and energy restriction (Experimental): Participants in this arm will consume 15% of energy as protein with 25% energy restriction.
  Interventions: Behavioral: Energy Restriction; Behavioral: Lower Protein

INTERVENTIONS:
Behavioral: Energy Restriction — Participants will receive an intervention specifically designed for adolescents and their group assignment that relies on nutrition education, nutritional counseling, social cognitive therapy, behavioral strategies, self-monitoring, portion size reduction, and increased physical activity.
  Participants will get an individualized dietary meal plan. Dietary counseling will be based on the MyPlate guidelines with extra attention and focus on appropriate protein food choice. Also in accordance to the MyPlate guidelines, all participants will be instructed to increase physical activity to 60 minutes a day as aerobic physical activity.
Behavioral: Higher protein — The higher protein group will be instructed to consume 30% of energy as protein, with 25% and 45% of energy from fat and carbohydrate, respectively.
  Arms: Higher protein and energy restriction
Behavioral: Lower Protein — The lower protein group will be instructed to consume 15% of energy as protein, with 25% and 60% of energy from fat and carbohydrate, respectively.
  Arms: Lower protein and energy restriction

SUMMARY:
The aim of the proposed study is to provide important data on weight loss efficacy in overweight and obese adolescents on an isocaloric higher protein diet vs a lower protein diet utilizing the U.S. Department of Agriculture (USDA) MyPlate nutrition guide. The investigators hypothesize that the higher protein diet will result in greater weight loss due to increased satiety and better dietary adherence.

DETAILED DESCRIPTION:
Aim 1 is to test the efficacy of a personalized higher protein weight loss intervention compared to a lower protein intervention which use the USDA MyPlate nutrition guide.

It is hypothesized that participants randomly assigned to the higher protein dietary treatment will lose more weight based on BMI-Z score over 12 weeks compared to participants in the lower dietary protein treatment.

Aim 2 is to test if changes in subjective ratings of appetite differ by dietary treatment (i.e. protein intake).

It is hypothesized that participants in the higher protein intervention will report a decrease in hunger and an increase in fullness compared to participants in the lower protein intervention.

Aim 3 is to test if change in the hexosamine biosynthetic pathway (HBP) measured at the rate limiting step of glutamine fructose-6-phosphate amidotransferase (GFAT) and glycosylation measured as O-linked N-acetylglucosamine (GlcNAc) transferase (OGT) differ by dietary treatment.

It is hypothesized that participants randomly assigned to the higher protein dietary treatment will have decreased change from baseline levels of GFAT and glycosylation (OGT) due to decreased carbohydrate intake compared to the lower protein treatment.

Exploratory Aims: As exploratory aims, the investigators will test if the higher protein or lower protein dietary treatments differentially alter glucose, insulin, cholesterol, and triglycerides (markers of the metabolic syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Be between the ages of 12 and 17, inclusive
* Be at or above the 85th BMI percentile (a number calculated from the participants height, weight, sex, and date of birth)
* Be willing to fast for 12 hours prior to clinic study visits 2 and 4
* Be willing to participate in the research study

Exclusion Criteria:

* Health Conditions:
* Has HIV or AIDS
* Has uncontrolled CVD or arrhythmia
* Has Type I or Type II diabetes.
* Is unable or unwilling to complete the study procedures
* Participant may not qualify for this study based on other exclusion criteria not listed. The study coordinator will go over this information in detail.

Medications:

* Diuretics
* Beta-blocker
* Weight loss medications, diet pills
* Anti-inflammatory drugs (corticosteroid/anabolic steroid/NSAID)
* Antipsychotic medications
* Other medications that may affect fluid balance or weight

Lifestyle:

• Plans to move out of the study area within the next 4 months, or plan to be out of the study area for more than 3 weeks during the course of the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
BMI Z-Score | up to Week 12

SECONDARY OUTCOMES:
Subjective Ratings of Appetite | Baseline and Week 12
Hexosamine Biosynthetic Pathway | Baseline and Week 12
  glutamine fructose-6-phosphate amidotransferase (GFAT) and glycosylation measured as O-linked N-acetylglucosamine (GlcNAc) transferase (OGT) measurement

OTHER OUTCOMES:
Glucose | Baseline and Week 12
Insulin | Baseline and Week 12
Cholesterol | Baseline and Week 12
Triglycerides | Baseline and Week 12
Blood Pressure | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States